CLINICAL TRIAL: NCT00271219
Title: Maternal Opioid Treatment: Human Experimental Research
Brief Title: RCT Comparing Methadone and Buprenorphine in Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hendree E. Jones, Professor, Dept of Psychiatry and Behavioral Sciences, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA15764-1; R01DA015764 (NIH); R01DA15764-1; DPMC
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-07

CONDITIONS: Opioid Related Disorders; Pregnancy; Opioid Dependence
Keywords: opiate addiction; opiate dependence; substance abuse; addiction; substance addiction; pregnancy; buprenorphine; methadone; fetal; neonatal; post-partum
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Methadone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Buprenorphine
  Interventions: Drug: Buprenorphine
- Methadone (Active Comparator): Methadone
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — daily oral dosing 20-140 mg
  Arms: Methadone
Drug: Buprenorphine — sl daily 2-32 mg
  Arms: Buprenorphine

SUMMARY:
Children born to women who abuse drugs have a high risk of being born with birth defects and developmental problems. Methadone is a drug that is commonly used for treating opioid dependence. However, its use by a pregnant woman can cause severe withdrawal symptoms in a newborn because of the prenatal exposure. The purpose of this study is to evaluate the effectiveness of buprenorphine, another drug, versus methadone in reducing withdrawal symptoms in children born to opioid-dependent women.

DETAILED DESCRIPTION:
Women who use drugs during pregnancy place their unborn children at high risk for being born addicted to drugs. Such children may also be born with birth defects and may experience learning and behavioral problems. Methadone, a synthetic narcotic, is commonly prescribed to treat opioid addiction. It may not be an optimal solution for opioid-dependent pregnant women, however, because a large percentage of children born to women taking methadone experience severe drug withdrawal symptoms at birth that often require medical treatment. Common opioid withdrawal symptoms, described as neonatal abstinence syndrome (NAS) in babies, include tremors, irritability, sleep problems, seizures, dehydration, and fever. Buprenorphine is a medication that has been approved to treat opioid dependence in individuals who are not pregnant but has not been approved for pregnant individuals. Past research has shown that use of buprenorphine in pregnant women results in improved birth outcomes over methadone. The purpose of this study is to evaluate the effectiveness of buprenorphine versus methadone at reducing opioid withdrawal symptoms in babies born to opioid-dependent women.

This study will enroll opioid-dependent pregnant women who are 13 to 30 weeks pregnant and will follow each woman and her child throughout the pregnancy until 6 weeks postpartum. All participants will undergo an initial screening that will last several hours. Participants will then be randomly assigned to receive either methadone or buprenorphine on a daily basis, and will be required to visit the clinic each day to receive their medication. Outcome measurements will be assessed at weekly study visits throughout the pregnancy, and will include drug use, HIV risk behaviors, medication dose adequacy and safety, treatment retention, and psychosocial functioning. Urine samples will be collected 3 times a week, and blood will be drawn throughout the pregnancy for safety monitoring. Outcome measurements related to the baby will include head circumference measurement, length of hospital stay, severity and frequency of withdrawal symptoms, and amount of medication needed to control withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence
* Current opioid use, as determined by a urine drug test
* Pregnant with a single child with a gestational age of 6 to 30 weeks, as determined by a sonogram

Exclusion Criteria:

* Current medical condition that would make study participation dangerous, as determined by study physician
* Diagnosed with an acute, severe psychiatric illness
* Current SCID I-E module diagnosis of benzodiazepine or alcohol abuse
* Use of alcohol or benzodiazepines in the 30 days prior to study entry, as determined by the Addiction Severity Index
* Pending legal action that may prohibit or interfere with study participation

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2005-07; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendree E. Jones, PhD, Principal Investigator — Johns Hopkins University
Locations (8):
- United States (6):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont
- Medical University of Vienna, Vienna, Austria
- St. Joseph's Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR. Nonserious adverse events in randomized trials with opioid-dependent pregnant women: direct versus indirect measurement. Am J Addict. 2012 Nov;21 Suppl 1:S1-4. doi: 10.1111/j.1521-0391.2012.00289.x. PMID 23786504
- [Derived] Holbrook AM, Jones HE, Heil SH, Martin PR, Stine SM, Fischer G, Coyle MG, Kaltenbach K. Induction of pregnant women onto opioid-agonist maintenance medication: an analysis of withdrawal symptoms and study retention. Drug Alcohol Depend. 2013 Sep 1;132(1-2):329-34. doi: 10.1016/j.drugalcdep.2013.02.031. Epub 2013 Mar 21. PMID 23523131
- [Derived] Jones HE, Heil SH, Tuten M, Chisolm MS, Foster JM, O'Grady KE, Kaltenbach K. Cigarette smoking in opioid-dependent pregnant women: neonatal and maternal outcomes. Drug Alcohol Depend. 2013 Aug 1;131(3):271-7. doi: 10.1016/j.drugalcdep.2012.11.019. Epub 2012 Dec 29. PMID 23279924
- [Derived] McNicholas LF, Holbrook AM, O'Grady KE, Jones HE, Coyle MG, Martin PR, Heil SH, Stine SM, Kaltenbach K. Effect of hepatitis C virus status on liver enzymes in opioid-dependent pregnant women maintained on opioid-agonist medication. Addiction. 2012 Nov;107 Suppl 1(0 1):91-7. doi: 10.1111/j.1360-0443.2012.04043.x. PMID 23106931
- [Derived] Holbrook AM, Baxter JK, Jones HE, Heil SH, Coyle MG, Martin PR, Stine SM, Kaltenbach K. Infections and obstetric outcomes in opioid-dependent pregnant women maintained on methadone or buprenorphine. Addiction. 2012 Nov;107 Suppl 1(Suppl 1):83-90. doi: 10.1111/j.1360-0443.2012.04042.x. PMID 23106930
- [Derived] Benningfield MM, Dietrich MS, Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Fischer G, Martin PR. Opioid dependence during pregnancy: relationships of anxiety and depression symptoms to treatment outcomes. Addiction. 2012 Nov;107 Suppl 1(0 1):74-82. doi: 10.1111/j.1360-0443.2012.04041.x. PMID 23106929
- [Derived] Coyle MG, Salisbury AL, Lester BM, Jones HE, Lin H, Graf-Rohrmeister K, Fischer G. Neonatal neurobehavior effects following buprenorphine versus methadone exposure. Addiction. 2012 Nov;107 Suppl 1(0 1):63-73. doi: 10.1111/j.1360-0443.2012.04040.x. PMID 23106928
- [Derived] Gaalema DE, Scott TL, Heil SH, Coyle MG, Kaltenbach K, Badger GJ, Arria AM, Stine SM, Martin PR, Jones HE. Differences in the profile of neonatal abstinence syndrome signs in methadone- versus buprenorphine-exposed neonates. Addiction. 2012 Nov;107 Suppl 1(0 1):53-62. doi: 10.1111/j.1360-0443.2012.04039.x. PMID 23106927
- [Derived] Kaltenbach K, Holbrook AM, Coyle MG, Heil SH, Salisbury AL, Stine SM, Martin PR, Jones HE. Predicting treatment for neonatal abstinence syndrome in infants born to women maintained on opioid agonist medication. Addiction. 2012 Nov;107 Suppl 1(0 1):45-52. doi: 10.1111/j.1360-0443.2012.04038.x. PMID 23106926
- [Derived] Salisbury AL, Coyle MG, O'Grady KE, Heil SH, Martin PR, Stine SM, Kaltenbach K, Weninger M, Jones HE. Fetal assessment before and after dosing with buprenorphine or methadone. Addiction. 2012 Nov;107 Suppl 1(0 1):36-44. doi: 10.1111/j.1360-0443.2012.04037.x. PMID 23106925
- [Derived] Jones HE, Fischer G, Heil SH, Kaltenbach K, Martin PR, Coyle MG, Selby P, Stine SM, O'Grady KE, Arria AM. Maternal Opioid Treatment: Human Experimental Research (MOTHER)--approach, issues and lessons learned. Addiction. 2012 Nov;107 Suppl 1(0 1):28-35. doi: 10.1111/j.1360-0443.2012.04036.x. PMID 23106924
- [Derived] Jones HE, Heil SH, Baewert A, Arria AM, Kaltenbach K, Martin PR, Coyle MG, Selby P, Stine SM, Fischer G. Buprenorphine treatment of opioid-dependent pregnant women: a comprehensive review. Addiction. 2012 Nov;107 Suppl 1(0 1):5-27. doi: 10.1111/j.1360-0443.2012.04035.x. PMID 23106923
- [Derived] Unger A, Jagsch R, Bawert A, Winklbaur B, Rohrmeister K, Martin PR, Coyle M, Fischer G. Are male neonates more vulnerable to neonatal abstinence syndrome than female neonates? Gend Med. 2011 Dec;8(6):355-64. doi: 10.1016/j.genm.2011.10.001. Epub 2011 Nov 15. PMID 22088886
- [Derived] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1074 Patients were screened for eligibility. 175 underwent randomization. 86 were assigned to receive buprenorphine. 58 of the patients assigned to buprenorphine completed the study. 89 were assigned to receive methadone. 73 of the patients assigned to methadone completed the study.
Pre-assignment Details: Of the 1074 screened: 243 did not give consent. 656 were excluded for a variety of reasons ranging from an estimated gestation age outside the range, to impending legal issues, to multiple-fetus pregnancy.
Groups:
- Methadone: Methadone
  Methadone : daily oral dosing 20-140 mg
- Buprenorphine: Buprenorphine
  Buprenorphine : sl daily 2-32 mg
Period: Overall Study
Arm/Group | Methadone | Buprenorphine
Started | 89 | 86
Completed | 73 | 58
Not Completed | 16 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Buprenorphine | Total
Number analyzed (Participants) | 73 | 58 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 58 | 131
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (0.7) | 25.3 (0.7) | 26.5 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 58 | 131
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 40 | 94
  Austria | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Child's Head Circumference Measurement (Measured at Birth)
Time Frame: birth
Measure: Mean (95% Confidence Interval); unit: cm
Groups:
- A Methadone: Methadone
  Methadone : daily oral dosing 20-140 mg
- B Buprenorphine: Buprenorphine
  Buprenorphine : sl daily 2-32 mg
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 73 | 58
cm | 33.0 [32.7 to 33.3] | 33.8 [33.5 to 34.1]

2. Primary Outcome: Child's Length of Hospital Stay
Time Frame: delivery until hospital discharge (min=2 days, max=79 days)
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 73 | 58
days | 17.5 [16 to 19] | 10.0 [8.8 to 11.2]

3. Primary Outcome: Number of Children Requiring Treatment for Neonatal Abstinence Signs (NAS)
Description: Neonatal abstinence syndrome (NAS) characterized by hyperirritability of the central nervous system and dysfunction in the autonomic nervous system, gastrointestinal tract, and respiratory system.11 When left untreated, NAS can result in serious illness (e.g., diarrhea, feeding difficulties, weight loss, and seizures) and death.
Time Frame: From birth until hospital discharge (min=4 days, max=10, depending on site)
Measure: Number; unit: participants
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 73 | 58
participants | 41 | 27

4. Primary Outcome: Child's Peak Daily Total NAS Score
Description: NAS was measured with the MOTHER NAS scale, which includes 28 items, 19 of which are used for scoring and medication decisions. Scores can range from 0 to 42, with higher scores indicating more severe withdrawal.
Time Frame: minimum twice daily from birth until NAS no longer measured (min=10 days)
Measure: Mean (95% Confidence Interval); unit: Score on the scale
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 73 | 58
Score on the scale | 12.8 [12.2 to 13.4] | 11.0 [10.4 to 11.6]

5. Primary Outcome: Total Amount of Morphine Sulfate That a Neonate Receives to Treat NAS
Description: Total amount in mg
Time Frame: Start of NAS treatment until discontinuation of NAS treatment (min=0 days, max=76 days)
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 73 | 58
mg | 10.4 [7.8 to 13] | 1.1 [0.4 to 1.8]

6. Secondary Outcome: Mother's Self-report of Drug Use (Measured Monthly by Time Line Follow Back)
Time Frame: monthly from study entry until discontinuation or delivery (min=29 days, max=239 days)
Population: frequency of use during the course of the study was too low to estimate the parameter with sufficient accuracy
Measure: Number; unit: percentage of drug use
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 89 | 86
percentage of drug use | NA — frequency of use during the course of the study was too low to estimate the parameter with sufficient accuracy | NA — frequency of use during the course of the study was too low to estimate the parameter with sufficient accuracy

7. Secondary Outcome: Mother's HIV Risk Behaviors (Measured Monthly by Risk Behavior Assessment)
Time Frame: monthly from study entry until discontinuation or delivery (min=29 days, max=239 days)
Population: frequency of occurrence too low to be estimated with accuracy
Measure: Number; unit: percentage of HIV risk behaviors
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 89 | 86
percentage of HIV risk behaviors | NA — frequency of occurrence too low to be estimated with accuracy | NA — frequency of occurrence too low to be estimated with accuracy

8. Secondary Outcome: Mother's Measures of Dose Adequacy and Acceptance Over Time (Measured Weekly by Dose Adequacy Measure)
Description: Pregnant women maintained on an opioid agonist medication may require upward adjustment to their medication during the course of pregnant. The Dose Adequacy Measure represented a recordation of dosing adjustments during the course of the study.
Time Frame: from study entry until discontinuation or delivery (min=29 days, max=239 days)
Population: intra-subject variability in dosing (typically 1 dose) over course of the trial was too small to estimate the parameter of interest with sufficient accuracy
Measure: Number; unit: dose increase per trimester
Arm/Group | A Methadone | B Buprenorphine
Number analyzed (Participants) | 89 | 86
dose increase per trimester | NA — intra-subject variability in dosing (typically 1 dose) over course of the trial was too small to estimate the parameter of interest with sufficient accuracy | NA — intra-subject variability in dosing (typically 1 dose) over course of the trial was too small to estimate the parameter of interest with sufficient accuracy

9. Secondary Outcome: Mother's Psychosocial Functioning at Delivery as Measured by the Addiction Severity Index Psychosocial Index Score
Description: The Addiction Severity Index is a structured clinical interview that assesses problem severity in 7 areas of functioning: alcohol use, drug use, medical, legal, employment, psychosocial, and psychiatric status. Each area of functioning yields a composite scale score between 0 and 1, with higher scores indicating greater problem severity in that area. Only the psychosocial index was examined in this study.
Time Frame: at delivery
Measure: Mean (95% Confidence Interval); unit: Score on the scale
Arm/Group | Methadone | Buprenorphine
Number analyzed (Participants) | 89 | 86
Score on the scale | .014 [-.134 to .166] | .088 [-.027 to .203]

ADVERSE EVENTS:
Time Frame: Entire course of the study, from baseline to end of study period (min=26 days, max=239 days)
Description: weekly assessment by self-report and clinician review with patient
Groups:
- Methadone: Mothers: Methadone
  Methadone : daily oral dosing 20-140 mg
- Buprenorphine: Mothers: Buprenorphine
  Buprenorphine : sl daily 2-32 mg
- Methadone: Neonates: Neonates born to mothers maintained on methadone
- Buprenorphine: Neonates: Neonates born to mothers maintained on buprenorphine
Arm/Group | Methadone: Mothers | Buprenorphine: Mothers | Methadone: Neonates | Buprenorphine: Neonates
Serious Adverse Events (participants affected / at risk) | 14/89 | 8/86 | 6/73 | 1/58
Other Adverse Events (participants affected / at risk) | 83/89 | 66/86 | 34/73 | 29/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Methadone: Mothers (N=89) | Buprenorphine: Mothers (N=86) | Methadone: Neonates (N=73) | Buprenorphine: Neonates (N=58)
Abnormal fetal health (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0/0 | 0/0 — Mothers only
cardiovascular (Cardiac disorders) | 1 | 0 | 2 | 1
gastrointestinal (Gastrointestinal disorders) | 1 | 1 | 0 | 1
genitourinary (Renal and urinary disorders) | 0 | 1 | 0 | 1
Illicit drug use (Psychiatric disorders) | 1 | 1 | 0/0 | 0/0 — Mothers only
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
neurological (Nervous system disorders) | 0 | 0 | 0 | 1
obstetrical (Pregnancy, puerperium and perinatal conditions) | 6 | 2 | 1 | 1
postsurgical (Surgical and medical procedures) | 0 | 0 | 0 | 1
psychological (Psychiatric disorders) | 1 | 0 | 0/0 | 0/0 — Mothers only
psychosocial (Social circumstances) | 1 | 0 | 0/0 | 0/0 — Mothers only
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
sexually transmitted diseases (Infections and infestations) | 1 | 0 | 0 | 0
skin conditions (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
sleep disturbances (Nervous system disorders) | 0 | 1 | 0/0 | 0/0 — Mothers only
other (General disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Methadone: Mothers (N=89) | Buprenorphine: Mothers (N=86) | Methadone: Neonates (N=73) | Buprenorphine: Neonates (N=58)
Abnormal fetal health (Pregnancy, puerperium and perinatal conditions) | 6 | 4 | 0/0 | 0/0 — Mothers only
abnormal appetite (Gastrointestinal disorders) | 2 | 0 | 4 | 1
abnormal laboratory values (General disorders) | 10 | 8 | 0 | 0
blood-borne disorders (Blood and lymphatic system disorders) | 5 | 1 | 0 | 1
cardiovascular (Cardiac disorders) | 29 | 14 | 8 | 4
endocrinologic (Endocrine disorders) | 5 | 3 | 1 | 1
eye, ear, nose, or throat problems (Ear and labyrinth disorders) | 12 | 15 | 1 | 1
fever (General disorders) | 3 | 2 | 0 | 0
gastrointestinal (Gastrointestinal disorders) | 60 | 47 | 5 | 4
genitourinary (Renal and urinary disorders) | 23 | 16 | 1 | 0
hematopoietic or lymphatic symptoms (Blood and lymphatic system disorders) | 14 | 15 | 17 | 14
Illicit drug use (Psychiatric disorders) | 10 | 8 | 3 | 5
dental problems (General disorders) | 22 | 15 | 1 | 2
musculoskeletal (Musculoskeletal and connective tissue disorders) | 38 | 28 | 3 | 1
neuromuscular (Nervous system disorders) | 33 | 29 | 0 | 0
neurological (Nervous system disorders) | 16 | 12 | 0 | 0
obstetrical (Pregnancy, puerperium and perinatal conditions) | 29 | 23 | 3 | 4
postsurgical (Surgical and medical procedures) | 16 | 8 | 3 | 0
psychological (Psychiatric disorders) | 24 | 21 | 0/0 | 0/0 — Mothers only
psychosocial (Social circumstances) | 4 | 5 | 0/0 | 0/0 — Mothers only
respiratory (Respiratory, thoracic and mediastinal disorders) | 29 | 31 | 14 | 12
sexually transmitted diseases (Infections and infestations) | 8 | 8 | 1 | 1
skin conditions (Skin and subcutaneous tissue disorders) | 16 | 12 | 7 | 2
sleep disturbances (Nervous system disorders) | 24 | 20 | 0/0 | 0/0 — Mothers only
somatic (Nervous system disorders) | 19 | 9 | 0/0 | 0/0 — Mothers only
other AE (General disorders) | 4 | 3 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes